CLINICAL TRIAL: NCT00813358
Title: Zenith TX2® TAA Endovascular Graft Post-approval Study
Brief Title: Zenith TX2® Post-market Approval Study
Acronym: TX2 2PAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-005; 370024, 2PAS
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Descending Thoracic Aortic Aneurysm
Keywords: Endovascular Aneurysm Repair; Aortic Aneurysm; Thoracic
MeSH Terms: conditions — Descending Thoracic Aortic Aneurysm; Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

ARMS (1):
- Endovascular repair (Experimental): treatment
  Interventions: Device: Zenith TX2® TAA Endovascular Graft

INTERVENTIONS:
Device: Zenith TX2® TAA Endovascular Graft — Endovascular treatment with the study device
  Other Names: TEVAR

SUMMARY:
The Zenith TX2® Post-market Approval Study is a clinical trial approved by US FDA to further study the safety and effectiveness of the Zenith TX2® TAA Endovascular Graft in the treatment of thoracic aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Descending thoracic aortic aneurysm with diameter greater than or equal to 5.0 cm; or
* Descending thoracic aortic aneurysm with a history of growth greater than or equal to 0.5 cm within the previous 12 months; or
* Descending thoracic aortic degenerative or atherosclerotic ulcers greater than or equal to 10 mm in depth and 20 mm in diameter

Exclusion Criteria:

* Age less than 18 years
* Other medical condition that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with limited life expectancy (i.e., less than 2 years)
* Pregnant, breast-feeding, or planning on becoming pregnant within 24 months
* Unwilling or unable to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Simultaneously participating in another investigative device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-07-10; Primary Completion 2020-02-14 (Actual); Study Completion 2020-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (24):
  - Kaiser Permanente, San Francisco, California
  - University of Denver Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Heart Care Midwest, Peoria, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Hospital of Queens, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - New York University, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - DFW Vascular Group, Dallas, Texas
  - Baylor University Medical Center at Dallas, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Harborview Medical Center, Seattle, Washington
- London Health Sciences Centre, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endovascular Repair
Started | 115
Completed | 46
Not Completed | 69
Not completed — Death | 32
Not completed — Lost to Follow-up | 12
Not completed — other endpoints | 5
Not completed — Withdrawal by Subject | 20

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 93
  Hispanic or Latino | 7
  Native Hawaiian - other Pacific Islander | 1
  Black or African Black or African American | 11
  Asian | 3
Region of Enrollment [Number; unit: participants]
  United States | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Thoracic Aortic Aneurysm-related Mortality
Description: Thoracic aortic aneurysm-related mortality defined as death from any cause occurring within 30 days of the initial procedure or a secondary intervention; or any death determined by the independent clinical events committee to be causally related to the initial implant procedure, secondary intervention, or rupture of the treated aneurysm.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Repair: Zenith® TX2® TAA Endovascular Graft through 5 years.
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 115
Participants | 114
Statistical Analysis 1: Comparison: Endovascular Repair; Test type: Non-Inferiority — NI=7%; KM product-limit estimator = 99.1, 95% CI 2-sided [97.4 to 100]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Endovascular Repair
All-Cause Mortality (participants affected / at risk) | 32/115
Serious Adverse Events (participants affected / at risk) | 83/115
Other Adverse Events (participants affected / at risk) | 14/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=115)
ANAEMIA (Blood and lymphatic system disorders) | 5 (6)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
CYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 4 (4)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3)
BRADYCARDIA (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 3 (3)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 (5)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 4 (4)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
CENTRAL NERVOUS SYSTEM EPIDERMOID TU (Congenital, familial and genetic disorders) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
VISION BLURRED (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
ENTEROCOLONIC FISTULA (Gastrointestinal disorders) | 1 (1)
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 (1)
FEMORAL HERNIA (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 8 (11)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2)
SPLENIC ARTERY ANEURYSM (Gastrointestinal disorders) | 1 (1)
ASTHENIA (General disorders) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1)
CHEST PAIN (General disorders) | 6 (6)
DEATH (General disorders) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 1 (1)
PHYSICAL DECONDITIONING (General disorders) | 1 (1)
PYREXIA (General disorders) | 2 (2)
STENT-GRAFT ENDOLEAK (General disorders) | 5 (5)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 2 (2)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1)
BACTEREMIA (Infections and infestations) | 2 (2)
CELLULITIS (Infections and infestations) | 2 (3)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1)
EPIDIDYMITIS (Infections and infestations) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 (1)
MENINGITIS (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 19 (19)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 8 (8)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 8 (12)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ARTERIAL BYPASS STENOSIS (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 3 (4)
INCOMPLETE SPINAL FUSION (Injury, poisoning and procedural complications) | 1 (1)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 (2)
BLOOD CREATININE INCREASE (Investigations) | 1 (1)
ENDOBRONCHIAL ULTRASOUND (Investigations) | 1 (1)
LABORATORY TEST ABNORMAL (Investigations) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
SACROILIAC JOINT DYSFUNCTION (Musculoskeletal and connective tissue disorders) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
CHRONIC MYELOID LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCOAST'S TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BRAIN INJURY (Nervous system disorders) | 1 (1)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 6 (7)
PARAPARESIS (Nervous system disorders) | 3 (3)
PARAPLEGIA (Nervous system disorders) | 4 (4)
SEIZURE (Nervous system disorders) | 1 (1)
SEIZURES (Nervous system disorders) | 1 (1)
SPINAL CORD ISCHAEMIA (Nervous system disorders) | 2 (2)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 (3)
DEVICE KINK (Product Issues) | 1 (1)
MEDICAL DEVICE ENTRAPMENT (Product Issues) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AORTO-BRONCHIAL FISTULA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHIAL SECRETION RETENTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEAS (Respiratory, thoracic and mediastinal disorders) | 5 (8)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (3)
CRANIOTOMY (Surgical and medical procedures) | 1 (1)
INCARCERATED HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
INTESTINAL RESECTION (Surgical and medical procedures) | 1 (1)
MECHANICAL VENTILATION (Surgical and medical procedures) | 5 (5)
OXYGEN THERAPY (Surgical and medical procedures) | 1 (1)
PANCREATECTOMY (Surgical and medical procedures) | 1 (1)
PERIPHERAL ENDARTERECTOMY (Surgical and medical procedures) | 1 (1)
PULMONARY RESECTION (Surgical and medical procedures) | 2 (2)
VASCULAR GRAFT (Surgical and medical procedures) | 1 (1)
ANEURYSM RUPTURED (Vascular disorders) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 3 (3)
AORTIC DISSECTION (Vascular disorders) | 2 (2)
AORTIC INTRAMURAL HAEMATOMA (Vascular disorders) | 1 (1)
ARTERIAL THROMBOSIS (Vascular disorders) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (4)
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY ANEURYSM RUPTURE (Vascular disorders) | 1 (1)
PERIPHERAL ARTERY OCCLUSION (Vascular disorders) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 2 (2)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1)
SUBCLAVIAN ARTERY OCCLUSION (Vascular disorders) | 2 (2)
THROMBOSIS (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (2)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
KNEE DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
KETONURIA (Renal and urinary disorders) | 1 (1)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (1)
RECTOCELE (Reproductive system and breast disorders) | 1 (1)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SPLENECTOMY (Surgical and medical procedures) | 1 (1)
ANEURYSM (Vascular disorders) | 1 (1)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=115)
ARRHYTHMIA (Cardiac disorders) | 6 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT00813358/Prot_SAP_000.pdf